CLINICAL TRIAL: NCT01080118
Title: A Clinical Trial on the Effectiveness of Video System in Improving Learning of Tracheal Intubation Using Standard Laryngoscopy Among Novices
Brief Title: Effectiveness of Video System in Improving Learning of Tracheal Intubation Using Standard Laryngoscopy Among Novices
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Gildasio De Oliveira, Gildasio De Oliveira, M.D. Principal Investigator, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: STU00007644
Record Dates: First submitted 2010-02-26; First posted 2010-03-03 (Estimated); Results first posted 2013-09-04 (Estimated); Last update posted 2013-12-02 (Estimated); Status verified 2013-10

CONDITIONS: Intubation Intraesophageal
Keywords: Teaching; Video Scope; Intubation
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- control group (Other): Control group, taught with a standard Macintosh laryngoscope
  Interventions: Other: Control group, taught with a standard Macintosh laryngoscope
- Study group (Experimental): Study group taught with the Airtraq video laryngoscope
  Interventions: Device: Airtraq

INTERVENTIONS:
Device: Airtraq — Subjects were taught with the Airtraq video laryngoscope
  Arms: Study group
Other: Control group, taught with a standard Macintosh laryngoscope — Subjects were taught how to use the Mackintosh blade first
  Arms: control group

SUMMARY:
The use of the video laryngoscope to teach laryngoscopy will improve the performance of tracheal intubation done by novices because it will allow a shared view of the airway leading to a better feedback from the trainer to the trainee.

DETAILED DESCRIPTION:
A group of 30 fourth year medical students and interns rotating through the department of anesthesiology will be studied. Firstly, a standard lecture will be provided in which the description and importance of laryngoscopy and tracheal intubation will be explained. This will include descriptions of anatomy, relevant equipment and technique of tracheal intubation. Following the lecture , the students will be randomly allocated using sealed envelopes into two groups : a control group ( taught with a standard Macintosh Laryngoscope ) and a study group ( taught with the Airtraq video laryngoscope).Each group will receive a demonstration and verbal instruction on how to perform laryngoscopy and tracheal intubation by their instructor.

ELIGIBILITY:
Students:

Inclusion criteria for the medical student:

* Medical student or intern rotating through the anesthesiology department

Exclusion criteria for the medical student:

* Previous attempts of laryngoscopy in humans
* Subject who refuses participation

Patients:

Inclusion Criteria:

* Age 18 -75 years of age
* ASA PS I, II
* Procedure that will require General anesthesia with tracheal intubation

Exclusion Criteria:

* Age < 18 years old or greater than 75 years of age
* Patient or student who refuses participation
* ASA Physical status class III or greater
* History of lung disease
* History of obstructive sleep apnea
* History of difficult intubation
* Evidence of possible difficult airway (Mallampati Class >2, TMH distance <6 cm, mouth opening <4 cm and limited neck mobility)
* Unanticipated difficult laryngoscopy (defined by inability of the attending anesthesiology to intubate after 2 attempts)
* Patients at risk for aspiration
* Patients with BMI greater than 35
* Pregnant patients

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2010-02; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gildasio DeOliveira, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern Memorial Hospital, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Medical students and intern trainees with no prior experience in laryngoscopy on clinical rotation in the Department of Anesthesiology were recruited to participate. Written informed consent was obtained from all the study participants.
Pre-assignment Details: Trainees received a structured lecture in airway management followed by training in laryngoscopy skills on a mannequin, and required to demonstrate proficiency. Trainees were then randomly assigned to attempt their first two intubations on different patients using either the optical or rigid laryngoscope with a MacIntosh size 3 blade.
Groups:
- Rigid Laryngoscope Group: Medical students or interns attempting intubation with standard size 3 Macintosh laryngoscope
- Video Laryngoscope Group: Medical students or interns attempting intubation with Airtraq video laryngoscope
- Rigid Laryngoscope Patients: Patients who were intubated using the rigid laryngoscope by the medical student of intern.
- Video Laryngoscope Patients: Patients who were intubated using the video laryngoscope by interns or medical student.
Period: Overall Study
Arm/Group | Rigid Laryngoscope Group | Video Laryngoscope Group | Rigid Laryngoscope Patients | Video Laryngoscope Patients
Started | 15 | 15 | 30 | 30
Completed | 15 | 15 | 30 | 30
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The 15 in each group represents the medical student/ interns who are being studied.
Groups:
- Total: Total of all reporting groups
Arm/Group | Rigid Laryngoscope Group | Video Laryngoscope Group | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 15 | 30
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 28 (3) | 27.5 (2) | 27.75 (2.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 11 | 12 | 23
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Successful Endotracheal Intubation
Description: A successful placement of the endotracheal tube as defined by the presence of bilateral breath sounds and positive recording of end tidal carbon dioxide.
Time Frame: 120 seconds
Population: The sample analysis was all of the medical students or interns who consented to participate in this study. All participants data was used for the analysis.
Measure: Number; unit: % successful
Arm/Group | Rigid Laryngoscope Group | Video Laryngoscope Group
Number analyzed (Participants) | 15 | 15
% successful | 33.3 | 83.3
Statistical Analysis 1: Comparison: Rigid Laryngoscope Group vs Video Laryngoscope Group; Test type: Superiority or Other; p = .001, t-test, 2 sided; Odds Ratio, log = .05, 99% CI 2-sided [.05 to .05]
Statistical Analysis 2: Comparison: Rigid Laryngoscope Group vs Video Laryngoscope Group; Test type: Non-Inferiority or Equivalence — Equivalence; p = .001, t-test, 2 sided

2. Secondary Outcome: Time to Intubation
Description: Time to intubation is the time interval of blade insertion until the removal of the laryngoscope.
Time Frame: 120 seconds
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: seconds
Arm/Group | Rigid Laryngoscope Group | Video Laryngoscope Group
Number analyzed (Participants) | 15 | 15
seconds | 75 [59 to 90] | 35 [27 to 44]

ADVERSE EVENTS:
Time Frame: 1 day
Arm/Group | Rigid Laryngoscope Group | Video Laryngoscope Group
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 9/15 | 1/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rigid Laryngoscope Group (N=15) | Video Laryngoscope Group (N=15)
mucosal laceration (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 1 (1) — Oral mucosa lacerated with introduction of device.

LIMITATIONS AND CAVEATS:
The intubating laryngeal mask airway the optical laryngoscope device used in this study does not allow for ventilation of the patient if intubation fails. We did not study retention of airway management skills between the groups.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No